CLINICAL TRIAL: NCT04038086
Title: Transport Von Peripheren Sättigungshormonen in Das Zentrale Nervensystem
Brief Title: Transport of Satiety Factors Into the CSF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 397/2019BO1
Record Dates: First submitted 2019-07-15; First posted 2019-07-30 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Glucose Tolerance Test; Circadian Rhythm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- oral glucose tolerance test (Experimental)
  Interventions: Diagnostic Test: oral glucose tolerance test
- circadian rhythm (Other)
  Interventions: Other: circadian rhythm
- effect of insulin on peptide transport (Experimental)
  Interventions: Drug: effect of insulin on peptide transport

INTERVENTIONS:
Diagnostic Test: oral glucose tolerance test — Participants will undergo an 75 gram oral glucose tolerance test. Blood and CSF will be collected in the fasting state before the test and every 30 minutes throughout the test which lasts for 2 hours.
  Arms: oral glucose tolerance test
Other: circadian rhythm — Blood and CSF will be collected five times throughout the day.
  Arms: circadian rhythm
Drug: effect of insulin on peptide transport — Blood and CSF will be collected in the fasting state and 15, 30, 60, 120 und 240 min after administration of 160 U of human insulin as nasal spray.
  Arms: effect of insulin on peptide transport

SUMMARY:
The blood-brain barrier regulates the passage of peripheral built appetite-suppressing hormones from the blood to the brain and informs the brain about the nutritional- and energy status.

The aim of this study is to investigate in which extent the hormones are able to overcome the blood-brain barrier and how long it takes after food intake. Relating thereto indications to the effect of peripheral hormones in the central nervous system and the role of these hormones in the development of overweight are provided.

In this study 30 patients (10 per intervention group) will be recruited. The patients are hospitalized in the local neurosurgery and they have a CSF-drainage due to their neurological primary disease or due to neurosurgical interventions. The patients are examined in each case on the same day.

Simultaneous samplings of blood and CSF are taken from 10 patients after an oral glucose tolerance test. These interventions are carried out to investigate in which extent the appetite-suppressing hormones (e.g. Leptin, Insulin, GLP 1 and Glucagon) reach the liquor and so the central nervous system.

In order to understand the temporal sequence, simultaneous samplings of blood and CSF are taken from 10 other patients at certain points throughout the day.

In a further group of 10 patients will be investigated how the central effective insulin modulates the transport of the other appetite-suppressing hormones. Therefore samplings of blood and CSF are investigated before and after intranasal insulin administration.

ELIGIBILITY:
Inclusion Criteria:

* patients with cerebrospinal fluid drainage

Exclusion Criteria:

* Women during pregnancy and lactation
* Participation in other interventional clinical trials
* severe infection within the last 4 months
* intake of central effective substances which may interact with the transport processes to be investigated
* hypersensitivity to any of the substances used
* diabetes mellitus
* Patients with CSF results indicative of infectious diseases within the central nervous system
* subjects with hemoglobin Hb <10 g / dl
* Patients with a neurosurgical disorder suspected of having a blood-brain barrier disorder

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-07-15 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Insulin transport into the CSF | Sample collection will be from 0 to 120 minutes in Arm 1, 18 hours in Arm 2, and 0 to 240 minutes in Arm 3
  Insulin will be measured in serum and CSF and the ratio will be calculated.

SECONDARY OUTCOMES:
Transport of proglucagon cleavage products into the CSF | Sample collection will be from 0 to 120 minutes in Arm 1, 18 hours in Arm 2, and 0 to 240 minutes in Arm 3
  Proglucagon cleavage products will be measured in serum and CSF and the ratio will be calculated.
Transport of FGF21 and FGF23 into the CSF | Sample collection will be from 0 to 120 minutes in Arm 1, 18 hours in Arm 2, and 0 to 240 minutes in Arm 3
  FGF21 and FGF23 will be measured in serum and CSF and the ratio will be calculated.
Ghrelin transport into the CSF | Sample collection will be from 0 to 120 minutes in Arm 1, 18 hours in Arm 2, and 0 to 240 minutes in Arm 3
  Ghrelin will be measured in serum and CSF and the ratio will be calculated.
PYY transport into the CSF | Sample collection will be from 0 to 120 minutes in Arm 1, 18 hours in Arm 2, and 0 to 240 minutes in Arm 3
  PYY will be measured in serum and CSF and the ratio will be calculated.
Leptin transport into the CSF | Sample collection will be from 0 to 120 minutes in Arm 1, 18 hours in Arm 2, and 0 to 240 minutes in Arm 3
  Leptin will be measured in serum and CSF and the ratio will be calculated.

OTHER OUTCOMES:
Association with hunger/satiety | fasting state (0 minutes) and last CSF collection (120 minutes in Arm 1, 18 hours in Arm 2, and 240 minutes in Arm 3)
  Association of the measured peptides with hunger/satiety ratings (assessed on a visual analog scale) will be tested.
Association with depression-like behaviour | fasting state (0 minutes) and last CSF collection (120 minutes in Arm 1, 18 hours in Arm 2, and 240 minutes in Arm 3)
  Association of the measured peptides with depression-like behaviour will be tested. Depression-like behaviour will be assessed by the BDI-II (Beck Depression Inventory) questionaire.
Association with mood | fasting state (0 minutes) and last CSF collection (120 minutes in Arm 1, 18 hours in Arm 2, and 240 minutes in Arm 3)
  Association of the measured peptides with mood will be tested. Mood will be assessed by PANAS (Positive and Negative Affect Schedule) questionaire.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Tuebingen, Department of Internal Medicine IV, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No
We will not be able to share patient level data due to data protection regulations.